CLINICAL TRIAL: NCT03241446
Title: A Phase I, Open-Label Study to Investigate the Pharmacokinetics and Dosimetry of Tc 99m Tilmanocept Following a Single Intravenous Dose Administration in Male and Female Subjects Diagnosed With Rheumatoid Arthritis
Brief Title: Pharmacokinetics and Dosimetry of Tc 99m Tilmanocept Following a Single Intravenous Dose Administration in Male and Female Subjects Diagnosed With Rheumatoid Arthritis (RA)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was combined with another trial that was on-going.
Sponsor: Navidea Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: NAV3-26
Record Dates: First submitted 2017-07-25; First posted 2017-08-07 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 50 ug Tilmanocept (Experimental): Single dose of 50 ug tilmanocept radiolabeled with 10 mCi technetium Tc99m
  Interventions: Drug: Tilmanocept
- 200 ug Tilmanocept (Experimental): Single dose of 200 ug tilmanocept radiolabeled with 10 mCi technetium Tc99m
  Interventions: Drug: Tilmanocept
- 400 ug Tilmanocept (Experimental): Single dose of 400 ug tilmanocept radiolabeled with 10 mCi technetium Tc99m
  Interventions: Drug: Tilmanocept

INTERVENTIONS:
Drug: Tilmanocept — Intravenously administered Technetium Tc 99m tilmanocept

SUMMARY:
A prospective, open-label, single center, study to evaluate pharmacokinetics and dosimetry of intravenously injected Tc 99m tilmanocept at three mass doses (50 µg, 200 µg, and 400 µg) radiolabeled with 10 millicuries (mCi) Tc 99m.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has provided written informed consent with HIPAA (Health Information Portability and Accountability Act) authorization before the initiation of any study-related procedures.
2. The subject is 30 - 65 years of age at the time of consent.
3. Has a negative urine drug screening for illicit or unprescribed drugs suggestive of drug abuse.
4. Subjects will have a BMI of 18 to 34 kg/m2, inclusive, at Screening
5. The subject has active RA as determined by the Clinical Disease Activity Index score of ≥ 10 and have ≥ 2 swollen joints.
6. If the subject is receiving methotrexate, they have been at a stable dose for > 4 weeks prior to the Day 1 visit.
7. If the subject is receiving biologic therapy or other DMARDs, they have been at a stable dose > 8 weeks prior to the Day 1 visit.
8. If the subject is receiving NSAIDS or oral corticosteroids, the dose has been at a stable dose for > 4 weeks prior to the Day 1 visit. The corticosteroid dose should be ≤ 10mg/day of prednisone or an equivalent steroid dose.
9. Aside from being diagnosed with rheumatoid arthritis, subjects must be in good health, as determined by medical history, physical examination, vital sign assessment, 12 lead electrocardiogram (ECG) and clinical laboratory evaluations.

Exclusion Criteria:

1. The subject is pregnant or lactating.
2. The subject has a significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder (as determined by the Investigator)
3. The subject has a history of significant hypersensitivity, intolerance, or allergy to dextran or modified forms of dextran; unless approved by the Investigator
4. The subject has a history or presence of an abnormal ECG, which, in the Investigator's opinion, is clinically significant
5. The subject has participated in a radiolabeled investigational study drug trial within 3 months prior to Day 1
6. The subject has exceeded yearly radioactive dose of 30 millisieverts (mSv)
7. The subject has a history of drug abuse or alcohol within 2 years before dose administration, or positive drug or alcohol test at screening.
8. The subject has used tobacco- or nicotine-containing products (including but not limited to cigarettes, e-cigarettes, pipes, cigars, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) within 6 months prior to Day 1, or positive cotinine screen
9. The subjects uses any prescription medications within 14 days prior to Day 1, except as allowed by the inclusion criteria or as deemed acceptable by the Investigator;
10. The subject uses any over-the-counter, non-prescription preparations (including vitamins, minerals, and phytotherapeutic/ herbal/plant-derived preparations) within 7 days prior to Day 1, unless deemed acceptable by the Investigator;
11. The subject has poor peripheral venous access;
12. The subject has donated blood within 30 days prior to Day 1, or plasma within 2 weeks prior to Day 1
13. The subject has received blood products within 2 months prior to Day 1;
14. The subject has any acute or chronic condition that, in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in this clinical study.
15. The subject has received any radiopharmaceutical within 7 days prior to the administration of Tc 99m tilmanocept.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09 (Estimated); Primary Completion 2018-01 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Maximum Plasma concentration (Cmax) of Technetium Tc 99m Tilmanocept | 1 Days
  Maximum Plasma concentration (Cmax) of Technetium Tc 99m Tilmanocept
Plasma Area Under the Curve (AUC) of Technetium Tc 99m Tilmanocept | 2 Days
  Plasma Area Under the Curve (AUC) of Technetium Tc 99m Tilmanocept
Systemic Clearance (CLs) of Technetium Tc 99m Tilmanocept | 3 Days
  Systemic Clearance (CLs) of Technetium Tc 99m Tilmanocept
Renal Clearance (CLr) of Technetium Tc 99m Tilmanocept | 2 days
  Renal Clearance (CLr) of Technetium Tc 99m Tilmanocept
Terminal Elimination Half-Life (T1/2) of Technetium Tc 99m Tilmanocept | 3 days
  Terminal Elimination Half-Life (T1/2) of Technetium Tc 99m Tilmanocept
Clinical Dosimetry of Technetium Tc 99m Tilmanocept | 3 days
  Clinical Dosimetry of Technetium Tc 99m Tilmanocept

SECONDARY OUTCOMES:
Incidence of Adverse Events | 7 Days
  Incidence of Adverse Events

IPD SHARING:
Plan to Share IPD: No